CLINICAL TRIAL: NCT01715038
Title: Home-fortification Approaches for the Prevention of Malnutrition in Pregnant and Lactating Women and Their Children in Bangladesh: Program Effectiveness Study
Brief Title: Effectiveness of LNS and MNP Supplements to Prevent Malnutrition in Women and Their Children in Bangladesh
Acronym: RDNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Family Health International 360 (Unknown); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); LAMB Project (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 252233; PR-10044 (Other: ICDDR,B)
Record Dates: First submitted 2012-10-18; First posted 2012-10-26 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Malnutrition
Keywords: malnutrition; stunting; LNS; micronutrient powder; hemoglobin
MeSH Terms: conditions — Malnutrition; Growth Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Comprehensive (Experimental): "Comprehensive" LNS: LNS-PLW provided daily to mothers during pregnancy and postpartum lactation (a total of at least 11 months, starting by 20 weeks gestation and ending at 6 months post-partum) and LNS developed for infants and young children (LNS-child) provided daily to their infants (beginning at 6 months of age for a period of 18 months i.e., from 6-24 months of age).
  Interventions: Dietary Supplement: LNS-PLW; Dietary Supplement: LNS-Child
- Child-only LNS (Experimental): "Child-only" LNS: Daily LNS-child supplementation of the child starting at 6 months of age and ending at 24 months of age (18 months total). Women will be provided with iron and folic acid (IFA) tablets during pregnancy and for 3 months postpartum.
  Interventions: Dietary Supplement: LNS-Child; Dietary Supplement: IFA
- Child-only MNP (Experimental): "Child-only" MNP: Daily MNP supplementation of the child starting at 6 months of age and ending at 24 months of age (18 months total). Women will be provided with iron and folic acid (IFA) tablets during pregnancy and for 3 months postpartum.
  Interventions: Dietary Supplement: MNP; Dietary Supplement: IFA
- Control: IFA (Active Comparator): Control: No additional nutrient supplementation for the child will be provided through the study, but the regular nutrition education and visits provided by the program frontline staff will continue. Women will be provided with iron and folic acid (IFA) tablets during pregnancy and for 3 months postpartum.
  Interventions: Dietary Supplement: IFA

INTERVENTIONS:
Dietary Supplement: LNS-PLW — Dietary supplement: Lipid-based nutrient supplement
  Lipid-based nutrient supplement for pregnant and lactating women (LNS-PLW)
  Daily dose of LNS-PLW will be 20 g, packaged in one sachet
  Arms: Comprehensive
Dietary Supplement: LNS-Child — Dietary supplement: Lipid-based nutrient supplement
  Lipid-based nutrient supplement for infants and young children (LNS-Child)
  Daily dose of LNS-Child will be 20 g, packaged in two 10 g sachets
  Arms: Child-only LNS; Comprehensive
Dietary Supplement: MNP — Dietary supplement: Micronutrient powder
  Micronutrient powder for infants and young children (MNP)
  The MNP for children will be packaged in 1 g sachets, so that each day, the child will consume one sachet.
  Arms: Child-only MNP
Dietary Supplement: IFA — Dietary supplement: Iron and folic acid nutrient supplement
  Iron-folic acid tablets for pregnant and lactating women
  Daily dose of iron-folic acid supplement will be one tablet containing 60 mg iron and 400 mcg folic acid
  Arms: Child-only LNS; Child-only MNP; Control: IFA

SUMMARY:
The program effectiveness study aims to assess the effect of a lipid-based nutrition supplement (LNS) and micronutrient powder (MNP) provided in a programmatic context for improving maternal nutritional status during pregnancy and lactation (LNS only), and preventing malnutrition in infants and young children (LNS and MNP) in Bangladesh.

DETAILED DESCRIPTION:
This study is a cluster-randomized controlled trial with four study "arms", implemented within the context of the Community Health and Development Program (CHDP) run by the World Mission Prayer League, which also has a hospital in the area and is known as LAMB. Data collection is longitudinal, starting with the identification of women in early pregnancy who are eligible to enter the study, and continuing, with follow-up of the child, until 24 months post-partum. A final follow-up visit will occur when the child is 36 months old to update contact information; no outcomes data will be collected at that final visit. The investigators are evaluating the effect of providing LNS-PLW to mothers during pregnancy and lactation on maternal health and nutrition outcomes (including anthropometric and micronutrient status), morbidity and birth outcomes in comparison to mothers who receive iron-folic acid tablets during pregnancy and lactation. The investigators are also evaluating the effect of three different home-fortification approaches (arms a-c, below) on child health and nutrition outcomes including anthropometric status, micronutrient status, anemia, and motor and cognitive development, in comparison to a control arm not receiving a home fortification intervention.

Additionally, the cost of implementation and delivery of the LNS-PLW, LNS-child or MNP interventions as part of the CHDP compared to standard CHDP program delivery will be documented. Willingness to pay (private demand) for LNS-PLW, LNS-child and MNP products by selected caregivers and male heads of households will be assessed at baseline and again at various points during the intervention period.

A process evaluation of the LNS and MNP interventions, and of the services provided to the control group, within the CHDP will be conducted to: 1) Document and evaluate the processes needed for implementation of interventions that provide a nutrient supplement such as LNS or MNP in the context of the CHDP; and 2) Explain and interpret program effectiveness study results and identify important facilitators and barriers to success of the nutrition intervention, which can be used to improve the effectiveness of current CHDP programs and future similar programs that include the scaling-up of LNS or MNP.

A post-intervention follow-up assessment for participants in the RDNS trial was added to the study protocol in November 2015. The intervention stopped when the study children turned 24 months old, and follow-up visits to update contact information were conducted when the children turned 36 months old. Thereafter, when the study children are between 40 and 52 months old, the follow-up assessment includes anthropometric and cognitive development assessments and collection of blood samples (finger prick, for measurement of hemoglobin) and buccal swab samples at the local clinics; for the mothers the follow-up includes anthropometric measurements, measurement of blood pressure and collection of fasting blood samples (finger prick). The follow-up also includes anthropometric measurements of the younger siblings, as well as a home visit to collect information on socioeconomic status, food security, hospitalizations of mother or child, developmental stimulation in the home, child food preferences and retrospective perceptions about the trial interventions.

Follow-up outcomes:

Maternal: Body mass index, skinfold thickness, mid-upper arm circumference, attained height. Hemoglobin, anemia, blood pressure, blood lipids, HbA1C.

Index child: Height, HAZ, stunting, weight, WHZ, WAZ, wasting, skinfold thickness, MUAC, arm fat and muscle area. Verbal ability (language), non-verbal ability (visual spatial), executive function and pre-academic skills. Hemoglobin, anemia. Hospitalizations since 24 months of age. Preferences for sweet and fatty foods.

Younger sibling: Height, HAZ, stunting, weight, WHZ, WAZ, wasting, MUAC.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≤ 20 weeks
* Planning to remain in the study area during pregnancy and the following three years (i.e., a permanent resident of the study area)

Exclusion Criteria:

* Pregnancy identified and registered in the CHDP program before the beginning of the enrollment.

Ages: 6 Months to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4011 (Actual)
Dates: Start 2011-10; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Birth weight | Within 48 hours (or back calculated from later measurements).
  Birth weight of the infants (women who received LNS-PLW vs. women who received iron-folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), time of year when outcome was assessed and child sex.
Birth length | Within 48 hours (or back calculated from later measurements)
  Birth length of the infants (women who received LNS-PLW vs. women who received iron-folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), time of year when outcome was assessed and child sex.
Child linear growth status at 24 months | 24 months
  Linear growth (the "comprehensive" LNS approach vs. the "child-only" LNS approach vs. "child-only" MNP) vis-à-vis one another and vis-à-vis the control group. Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), time of year when outcome was assessed and child sex.

SECONDARY OUTCOMES:
Change in maternal weight between baseline and 36 wk gestation | Between 12-20 and 36 weeks of gestation
  Gestational weight gain from enrollment (by 20 weeks of gestation) through 36 weeks of gestation (women who received LNS for pregnant and lactating women (LNS-PLW) vs. a comparison group who received the standard care, iron-folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment) and time of year when outcome was assessed.
Pre-eclampsia | 36 weeks of gestation
  Prevalence of pre-eclampsia (women who received LNS-PLW vs. women who received iron and folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment) and time of year when outcome was assessed.
Duration of gestation | Day 0
  Duration of gestation (women who received LNS-PLW vs. women who received iron and folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment) and time of year when outcome was assessed.
Pre-term delivery | Day 0
  Prevalence of pre-term delivery (delivery at <37 gestational weeks) in the infants (women who received LNS-PLW vs. women who received iron-folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), time of year when outcome was assessed and child sex.
Low birth weight | Within 48 hours (or back calculated from later measurements)
  Prevalence of low birth weight (birth weight < 2500 g) in the infants (women who received LNS-PLW vs. women who received iron-folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), time of year when outcome was assessed and child sex.
Small for gestational age (SGA) | Within 48 hours (or back calculated from later measurements)
  Prevalence of SGA (birth weight < 10th percentile) in the infants (women who received LNS-PLW vs. women who received iron-folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), time of year when outcome was assessed and child sex.
Newborn stunting | Within 48 hours (or back calculated from later measurements)
  Prevalence of newborn stunting (length-for-age z-score <-2) in the infants (women who received LNS-PLW vs. women who received iron-folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), time of year when outcome was assessed and child sex.
BMI z score at birth | Within 48 hours (or back calculated from later measurements)
  BMI z score at birth (women who received LNS-PLW vs. women who received iron-folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), time of year when outcome was assessed and child sex.
Head circumference (HC) at birth | Within 48 hours (or back calculated from later measurements)
  Head circumference at birth of the infants (women who received LNS-PLW vs. women who received iron-folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), time of year when outcome was assessed and child sex.
Small head size at birth | Within 48 hours (or back calculated from later measurements)
  Prevalence of small head size (HC-z-score <-2) at birth (women who received LNS-PLW vs. women who received iron-folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), time of year when outcome was assessed and child sex.
Change in maternal weight between 42 d and 6 mo postpartum | Between 42 d and 6 mo postpartum
  Postpartum weight change from 42 days through 6 mo postpartum (women who received LNS for pregnant and lactating women (LNS-PLW) vs. a comparison group who received the standard care, iron-folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), for time of year when outcome was assessed
Change in maternal iodine status between baseline and 6 mo postpartum | Between 10-20 weeks of gestation and 6 months postpartum
  Prevalence of iodine deficiency during lactation (women who received LNS-PLW vs. women who received iron and folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal iodine status, baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment) and time of year when outcome was assessed.
Change in maternal iron status between baseline and 6 months postpartum | Between 10-20 weeks of gestation and 6 months postpartum
  Prevalence of iron deficiency during lactation (women who received LNS-PLW vs. women who received iron and folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal iron status, baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment) and time of year when outcome was assessed.
Change in maternal iron-deficiency anemia between baseline and 6 months postpartum | Between 10-20 weeks of gestation and 6 months postpartum
  Prevalence of iron-deficiency anemia during lactation (women who received LNS-PLW vs. women who received iron and folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal iron status, baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment) and time of year when outcome was assessed.
Change in maternal anemia between baseline and 6 months postpartum | Between 10-20 weeks of gestation and 6 months postpartum
  Prevalence of anemia during lactation (women who received LNS-PLW vs. women who received iron and folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal anemia status, baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment) and time of year when outcome was assessed.
Change in maternal vitamin A status between baseline and 6 months postpartum | Between 10-20 weeks of gestation and 6 months postpartum
  Prevalence of vitamin A deficiency during lactation (women who received LNS-PLW vs. women who received iron and folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal vitamin A status, baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment) and time of year when outcome was assessed.
Change in maternal depressive symptoms between baseline and 6 months postpartum | Between 10-20 weeks of gestation and 6 months postpartum
  Prevalence of depression during lactation (women who received LNS-PLW vs. a comparison group). Pre-defined tests for interaction will be done for: baseline maternal depression status, baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment) and time of year when outcome was assessed.
Child hemoglobin concentration at 18 months of age | 18 months
  Hemoglobin concentration (the "comprehensive" LNS approach vs. the "child-only" LNS approach vs. "child-only" MNP) vis-à-vis one another and vis-à-vis the control group. Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), time of year when outcome was assessed and child sex.
Child iron status at 18 months of age | 18 months
  Prevalence of iron deficiency (the "comprehensive" LNS approach vs. the "child-only" LNS approach vs. "child-only" MNP) vis-à-vis one another and vis-à-vis the control group. Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), time of year when outcome was assessed and child sex.
Child vitamin A status at 18 months of age | 18 months
  Prevalence of vitamin A deficiency (the "comprehensive" LNS approach vs. the "child-only" LNS approach vs. "child-only" MNP) vis-à-vis one another and vis-à-vis the control group. Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), time of year when outcome was assessed and child sex.
Child anemia status at 18 months of age | 18 months
  Prevalence of anemia in children (the "comprehensive" LNS approach vs. the "child-only" LNS approach vs. "child-only" MNP) vis-à-vis one another and vis-à-vis the control group. Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), time of year when outcome was assessed and child sex.
Child iron-deficiency anemia status at 18 months of age | 18 months
  Prevalence of iron-deficiency anemia in children (the "comprehensive" LNS approach vs. the "child-only" LNS approach vs. "child-only" MNP) vis-à-vis one another and vis-à-vis the control group. Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), time of year when outcome was assessed and child sex.
Wasting at 24 months of age | 24 months
  Prevalence of wasting (weight-for-length z-score <-2) in children (the "comprehensive" LNS approach vs. the "child-only" LNS approach vs. "child-only" MNP) vis-à-vis one another and vis-à-vis the control group. Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), time of year when outcome was assessed and child sex.
Head circumference at 24 months of age | 24 months
  Head circumference of children (the "comprehensive" LNS approach vs. the "child-only" LNS approach vs. "child-only" MNP) vis-à-vis one another and vis-à-vis the control group. Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), time of year when outcome was assessed and child sex.
Stunting at 24 months of age | 24 months
  Prevalence of stunting (length-for-age z-score <-2) in children (the "comprehensive" LNS approach vs. the "child-only" LNS approach vs. "child-only" MNP) vis-à-vis one another and vis-à-vis the control group. Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), time of year when outcome was assessed and child sex.
Child motor development at 24 months of age | 24 months
  Motor development of children (the "comprehensive" LNS approach vs. the "child-only" LNS approach vs. "child-only" MNP) vis-à-vis one another and vis-à-vis the control group. Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), time of year when outcome was assessed and child sex.
Child cognitive development at 24 months of age | 24 months
  Cognitive development of children (the "comprehensive" LNS approach vs. the "child-only" LNS approach vs. "child-only" MNP) vis-à-vis one another and vis-à-vis the control group. Pre-defined tests for interaction will be done for: baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment), time of year when outcome was assessed and child sex.

OTHER OUTCOMES:
Change in maternal hemoglobin concentration between baseline and 36 wk gestation | Between 12-20 weeks and 36 weeks of gestation
  Hemoglobin concentration during pregnancy (women who received LNS-PLW vs. women who received iron-folic acid tablets). Pre-defined tests for interaction will be done for: hemoglobin baseline value, baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment) and time of year when outcome was assessed.
Change in maternal iodine status between baseline and 36 wk gestation | Between 12-20 weeks and 36 weeks of gestation
  Prevalence of iodine deficiency during pregnancy (women who received LNS-PLW vs. women who received iron and folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal iodine status, baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment) and time of year when outcome was assessed.
Change in maternal depressive symptoms between baseline and 36 wk gestation | Between 12-20 weeks and 36 weeks of gestation
  Prevalence of depression during pregnancy (women who received LNS-PLW vs. a comparison group). Pre-defined tests for interaction will be done for: baseline maternal depression status, baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment) and time of year when outcome was assessed.
Change in maternal iron status between baseline and 36 wk gestation | Between 12-20 weeks and 36 weeks of gestation
  Prevalence of iron deficiency during pregnancy (women who received LNS-PLW vs. women who received iron and folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal iron status, baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment) and time of year when outcome was assessed.
Change in maternal vitamin A status between baseline and 36 wk gestation | Between 12-20 weeks and 36 weeks of gestation
  Prevalence of vitamin A deficiency during pregnancy (women who received LNS-PLW vs. women who received iron and folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal vitamin A status, baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment) and time of year when outcome was assessed.
Change in maternal anemia between baseline and 36 wk gestation | Between 12-20 weeks and 36 weeks of gestation
  Prevalence of anemia during pregnancy (women who received LNS-PLW vs. women who received iron and folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal anemia status, baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment) and time of year when outcome was assessed.
Change in maternal iron-deficiency anemia between baseline and 36 wk gestation | Between 12-20 weeks and 36 weeks of gestation
  Prevalence of iron-deficiency anemia during pregnancy (women who received LNS-PLW vs. women who received iron and folic acid tablets). Pre-defined tests for interaction will be done for: baseline maternal iron-deficiency anemia status, baseline maternal characteristics (age, height, BMI, education, primiparity, food insecurity, wealth and gestational age at enrollment) and time of year when outcome was assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn G Dewey, PhD, Principal Investigator — University of California, Davis
Locations (1):
- LAMB, Parbatipur, Rangpur and Dinajpur Districts, Bangladesh

REFERENCES:
- [Derived] Roy A, Hossain MM, Ullah MB, Mridha MK. Maternal and neonatal peripartum factors associated with late initiation of breast feeding in Bangladesh: a secondary analysis. BMJ Open. 2022 May 18;12(5):e051004. doi: 10.1136/bmjopen-2021-051004. PMID 35584874
- [Derived] Ullah MB, Mridha MK, Arnold CD, Matias SL, Khan MSA, Siddiqui Z, Hossain M, Paul RR, Dewey KG. Factors associated with diarrhea and acute respiratory infection in children under two years of age in rural Bangladesh. BMC Pediatr. 2019 Oct 27;19(1):386. doi: 10.1186/s12887-019-1738-6. PMID 31656181
- [Derived] Ullah MB, Mridha MK, Arnold CD, Matias SL, Khan MSA, Siddiqui Z, Hossain M, Dewey KG. Provision of Pre- and Postnatal Nutritional Supplements Generally Did Not Increase or Decrease Common Childhood Illnesses in Bangladesh: A Cluster-Randomized Effectiveness Trial. J Nutr. 2019 Jul 1;149(7):1271-1281. doi: 10.1093/jn/nxz059. PMID 31162588
- [Derived] Matias SL, Mridha MK, Young RT, Hussain S, Dewey KG. Daily Maternal Lipid-Based Nutrient Supplementation with 20 mg Iron, Compared with Iron and Folic Acid with 60 mg Iron, Resulted in Lower Iron Status in Late Pregnancy but Not at 6 Months Postpartum in Either the Mothers or Their Infants in Bangladesh. J Nutr. 2018 Oct 1;148(10):1615-1624. doi: 10.1093/jn/nxy161. PMID 30204885
- [Derived] Matias SL, Mridha MK, Young RT, Khan MSA, Siddiqui Z, Ullah MB, Vosti SA, Dewey KG. Prenatal and Postnatal Supplementation with Lipid-Based Nutrient Supplements Reduces Anemia and Iron Deficiency in 18-Month-Old Bangladeshi Children: A Cluster-Randomized Effectiveness Trial. J Nutr. 2018 Jul 1;148(7):1167-1176. doi: 10.1093/jn/nxy078. PMID 29901736
- [Derived] Adams KP, Ayifah E, Phiri TE, Mridha MK, Adu-Afarwuah S, Arimond M, Arnold CD, Cummins J, Hussain S, Kumwenda C, Matias SL, Ashorn U, Lartey A, Maleta KM, Vosti SA, Dewey KG. Maternal and Child Supplementation with Lipid-Based Nutrient Supplements, but Not Child Supplementation Alone, Decreases Self-Reported Household Food Insecurity in Some Settings. J Nutr. 2017 Dec;147(12):2309-2318. doi: 10.3945/jn.117.257386. Epub 2017 Oct 4. PMID 28978680
- [Derived] Mridha MK, Matias SL, Paul RR, Hussain S, Sarker M, Hossain M, Peerson JM, Vosti SA, Dewey KG. Prenatal Lipid-Based Nutrient Supplements Do Not Affect Pregnancy or Childbirth Complications or Cesarean Delivery in Bangladesh: A Cluster-Randomized Controlled Effectiveness Trial. J Nutr. 2017 Sep;147(9):1776-1784. doi: 10.3945/jn.117.248880. Epub 2017 Jul 19. PMID 28724657
- [Derived] Mridha MK, Matias SL, Paul RR, Hussain S, Khan MSA, Siddiqui Z, Ullah B, Sarker M, Hossain M, Young RT, Arnold CD, Dewey KG. Daily Consumption of Lipid-Based Nutrient Supplements Containing 250 mug Iodine Does Not Increase Urinary Iodine Concentrations in Pregnant and Postpartum Women in Bangladesh. J Nutr. 2017 Aug;147(8):1586-1592. doi: 10.3945/jn.117.248963. Epub 2017 Jun 14. PMID 28615379
- [Derived] Matias SL, Mridha MK, Tofail F, Arnold CD, Khan MS, Siddiqui Z, Ullah MB, Dewey KG. Home fortification during the first 1000 d improves child development in Bangladesh: a cluster-randomized effectiveness trial. Am J Clin Nutr. 2017 Apr;105(4):958-969. doi: 10.3945/ajcn.116.150318. Epub 2017 Mar 8. PMID 28275128
- [Derived] Dewey KG, Mridha MK, Matias SL, Arnold CD, Cummins JR, Khan MS, Maalouf-Manasseh Z, Siddiqui Z, Ullah MB, Vosti SA. Lipid-based nutrient supplementation in the first 1000 d improves child growth in Bangladesh: a cluster-randomized effectiveness trial. Am J Clin Nutr. 2017 Apr;105(4):944-957. doi: 10.3945/ajcn.116.147942. Epub 2017 Mar 8. PMID 28275125
- [Derived] Matias SL, Mridha MK, Paul RR, Hussain S, Vosti SA, Arnold CD, Dewey KG. Prenatal Lipid-Based Nutrient Supplements Affect Maternal Anthropometric Indicators Only in Certain Subgroups of Rural Bangladeshi Women. J Nutr. 2016 Sep;146(9):1775-82. doi: 10.3945/jn.116.232181. Epub 2016 Jul 20. PMID 27440259
- [Derived] Harding KL, Matias SL, Mridha MK, Moniruzzaman M, Vosti SA, Hussain S, Dewey KG, Stewart CP. Adherence to recommendations on lipid-based nutrient supplement and iron and folic acid tablet consumption among pregnant and lactating women participating in a community health programme in northwest Bangladesh. Matern Child Nutr. 2017 Jan;13(1):e12252. doi: 10.1111/mcn.12252. Epub 2016 Feb 22. PMID 26898720
- [Derived] Mridha MK, Matias SL, Chaparro CM, Paul RR, Hussain S, Vosti SA, Harding KL, Cummins JR, Day LT, Saha SL, Peerson JM, Dewey KG. Lipid-based nutrient supplements for pregnant women reduce newborn stunting in a cluster-randomized controlled effectiveness trial in Bangladesh. Am J Clin Nutr. 2016 Jan;103(1):236-49. doi: 10.3945/ajcn.115.111336. Epub 2015 Nov 25. PMID 26607935